CLINICAL TRIAL: NCT04422366
Title: A Multicenter,Randomized,Blind and Positive-Controlled Phase Ⅲ Study to Evaluate the Efficacy, Immunogenicity and Safety of the 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 20-45 Years
Brief Title: Evaluate the Efficacy, Immunogenicity and Safety of 9-valent HPV Recombinant Vaccine in Chinese Healthy Females
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9-HPV-3001
Record Dates: First submitted 2020-05-17; First posted 2020-06-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; CIN1; CIN2; CIN3; VaIN1; VaIN2; VaIN3; Genital Wart; VIN 1; VIN 2; VIN 3; AIS
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata | interventions — Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 (Experimental): Participants in this arm would receive 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha)
  Interventions: Biological: 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha)
- GARDASIL® (Active Comparator): Participants in this arm would receive GARDASIL®
  Interventions: Biological: GARDASIL®

INTERVENTIONS:
Biological: 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) — Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule.
  Arms: 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52
Biological: GARDASIL® — Subjects received 3 doses of Placebo according to a 0, 2, 6-month schedule
  Arms: GARDASIL®

SUMMARY:
This study is designed to evaluate the vaccine efficacy, immunogenicity and safety of the 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 20-45 Years .

ELIGIBILITY:
Inclusion Criteria:

(If the "*" option is not met during screening, the visit can be rescheduled)

* Chinese women aged 20-45 who can provide legal identification and have a sexual life history;
* The subject fully understands the study procedures, understands the risks and benefits associated with participating in the study, and voluntarily signs the informed consent;
* Subjects are able to read, understand and fill in application forms such as diary CARDS and contact CARDS, and participate in follow-up according to the study requirements;
* Subjects have not been screened for cervical cancer, or have been screened for cervical cancer but the results are normal;
* *0 days before the gynecological visit, no sex within 48 hours, no flushing or vaginal cleaning within 72 hours, no use of vaginal drugs or preparations;Subject agrees to refrain from sexual intercourse (including anal, vaginal, or genital/genital contact of the same or opposite sex) for 48 hours prior to any visit that includes gynecological sample collection, and to refrain from vaginal flushing, vaginal cleansing, or use of vaginal medications or preparations for 72 hours;
* When the subjects were enrolled, the urine pregnancy test was negative (sensitivity was 25mIU/ml cox-hcg), they were not in the lactation period and had no family planning within 7 months after enrollment (1 month before whole-course inoculation).2 weeks before included in the study, effective contraceptive measures has been adopted and agreed to in the first seven months after the study (vaccinations after 1 months ago) continue to adopt effective contraceptive measures (effective contraceptive measures include: the pill, injection or embedded contraception, slow-release local birth control pills, hormone patch, the intrauterine device (IUD), sterilization, abstinence, condom (men), diaphragm, cervical cap, etc.), rhythm, withdrawal and emergency contraception is unacceptable contraception;
* *body temperature <37.3℃ (underarm body temperature)

Exclusion Criteria:

First dose exclusion criteria(If the "*" option is met during screening, the visit can be rescheduled)

* Have been vaccinated with commercially available HPV vaccine in the past or planned to be vaccinated with commercially available HPV vaccine during the study period;Or have participated in a clinical trial of the HPV vaccine and have received a vaccine/placebo vaccination;
* Previous positive history of HPV;
* Has a history of abnormal cervical cytology, including squamous intraepithelial lesions (SIL) or not clear meaning of the atypical squamous cells (ASC - US), except the atypical squamous cells - not highly squamous intraepithelial lesion (ASC - H), atypical glandular epithelial cells, or those with cervical intraepithelial neoplasia (CIN) and carcinoma in situ or abnormal cervical biopsy results such as the history;
* Past history of anal and genital diseases (such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, vulvar cancer, vaginal cancer and anal cancer, etc.);
* Received total hysterectomy or pelvic radiotherapy;
* Cervical insufficiency or abnormal cervical structure (judged by the results of routine gynecological examination);
* Previous sexual history (including syphilis, gonorrhea, chancre, venereal lymphatic granuloma, granuloma inguinal) or have obvious condyloma;
* A history of seizures, convulsions or convulsions, or a family history of mental illness;
* Have participated in other gynecology-related clinical trials within 6 months, and have used or plan to use other investigational or unregistered products (drugs or vaccines) other than the vaccine in this study within 3 months;
* A history of severe allergies requiring medical intervention, such as anaphylactic shock, anaphylactic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.A history of severe adverse reactions to previous vaccinations or a history of severe allergies to any of the components of the vaccine under study (histidine, polysorbate, aluminum phosphate, sodium borate, amorphous aluminum phosphate sulfate adjuvant and water for injection) (such as swelling of the mouth and throat, dyspnea, hypotension or shock, severe urticaria, etc.);
* Subject receives any immunoglobulin or blood product within 3 months prior to the first dose of vaccination, or plans to receive such product within the next 7 months (1 month prior to the full course of vaccination);
* Subjects present/present with immune impairment or have been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases;
* Immunosuppressant therapy within 1 month before the first dose of vaccination, such as long-term use of systemic glucocorticoid therapy (≥2mg/kg/ day, for more than 2 weeks, such as prednisone or similar drugs;Topical administration (such as ointment, eye drops, inhalant or nasal spray) not exceeding the recommended dosage in the directions or showing any signs of systemic exposure) or planning to receive such treatment within the next 7 months (1 month before the full course of inoculation);
* Absence of spleen or functional absence of spleen, and absence of spleen or splenectomy in any case;
* Patients with severe liver, kidney and cardiovascular diseases, diabetes or malignant tumor with complications;
* Patients with thrombocytopenia or any coagulation disorders that may be contraindications to intramuscular injection;
* * subjects received inactivated or recombinant vaccines within 14 days prior to study enrollment, or attenuated live vaccines within 28 days prior to study enrollment;
* * an acute illness or an acute episode of a chronic illness within 3 days prior to vaccination or the use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
* * the first dose of vaccine was in pregnancy at the time of vaccination, or the end of pregnancy had not exceeded 6 weeks;
* * after questioning, subjects had fever symptoms (subaxillary body temperature ≥37.3℃) before the first day of vaccination (within 24 hours before vaccination);
* * the subject is in the menstrual period;
* * severe acute vaginitis and suppurative cervicitis found by naked eye during gynecological examination (purulent secretion visible by naked eye);
* Blood pressure on physical examination before the first dose of vaccination was higher than normal or increased (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg);
* Gynecological examination before the first dose of vaccination suspected genital warts, or on the basis of clinical symptoms and signs suspected vulva, vagina or cervical precancerous lesions and the possibility of cancer;
* Subjects may be unable to comply with the study procedure, comply with the agreement, or plan to permanently relocate from the region prior to completion of the study, or may be permanently absent from the region during the scheduled visit;
* In the opinion of the investigators, the subjects had any other factors that made them unsuitable to participate in the clinical trial, so that continued participation in the study could not guarantee the maximum benefit of the subjects.

Second and third doses of vaccine were excluded criteria

* new discoveries or new occurrences that meet the first dose exclusion criteria (except for articles 2, 3, 4, 21);
* other serious adverse events: the investigator decides whether to terminate the experimental vaccination according to its treatment needs;
* the investigator assays for any other reasons that may be considered necessary to terminate the trial vaccination.

Second and third doses of vaccine were delayed criteria

Vaccination may be postponed if:

* fever (underarm body temperature ≥37.3℃);
* before inoculation (on the day of inoculation), the urine pregnancy test was positive (sensitivity was 25mIU/ml n-hcg);
* acute illness or acute attack of a chronic disease or use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days before vaccination;
* insufficient interval between other vaccines (inactivated or recombinant vaccines received within 14 days prior to vaccination, or any live attenuated vaccine received within 28 days);
* any immunoglobulin or blood products received during vaccination should be administered at least 3 months after the vaccination;
* other circumstances that can be postponed as judged by the researcher.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8000 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related high-grade cervical abnormalities (CIN 2/3) at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84

SECONDARY OUTCOMES:
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related 6-month and 12-month Persistent Infection at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related VIN 1/2/3, VaIN1/2/3, AIN1/2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related VIN 2/3, VaIN2/3, AIN2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of other HPV types related CIN 2/3 at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of other HPV types related VIN 1/2/3, VaIN1/2/3, AIN1/2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related high-grade cervical abnormalities (CIN 2/3) at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related 6-month and 12-month Persistent Infection at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related VIN 2/3, VaIN2/3, AIN2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of HPV 31-, 33-, 45-, 52-, and 58-related VIN 1/2/3, VaIN1/2/3, AIN1/2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of other HPV types related VIN 2/3, VaIN2/3, AIN2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 3 | 1 month post vaccination 3 (Month 7) up to Month 84
The person-year incidence of other HPV types related CIN 2/3 at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of other HPV types related VIN 1/2/3, VaIN1/2/3, AIN1/2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
The person-year incidence of other HPV types related VIN 2/3, VaIN2/3, AIN2/3, vulvar cancer, vaginal cancer and anal cancer at least 1 month post Dose 1 | 1 month post vaccination 1 up to Month 84
Percentage of Participants Who Report at Least 1 Solicited Injection-site and Systemic Adverse Event 30 minutes post any vaccination | 30 minutes post any vaccination
Percentage of Participants Who Report at Least 1 Solicited Adverse Event 7 days post any vaccination | 7 days post any vaccination
Percentage of Participants Who Report at Least 1 Solicited and Unsolicited Adverse Event 30 days post any vaccination | 30 days post any vaccination
Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) from 1st vaccination to the completion of study | 1 month post vaccination 3 (Month 7) up to Month 84
Percentage of Participants Who Experience Pregnancy from 1st vaccination to the completion of study | 1 month post vaccination 3 (Month 7) up to Month 84
neutralizing antibody level | 30 days post third dose of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Liuzhou center for disease control and prevention, Liuchow, Guangxi, China